CLINICAL TRIAL: NCT06514846
Title: Utilizing the Michigan Neuropathy Screening Instrument, Routine Nerve Conduction Study (NCS), and Nerve Ultrasound for Early Detection of Diabetic Neuropathy
Brief Title: Utilizing the Michigan Neuropathy Screening Instrument for Early Detection of Diabetic Neuropathy
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Reda Khalafallah Khalil, Principal investigator, Sohag University
Other Study IDs: Soh-Med-24-06-01MS
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Polyneuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients Group: Study Population:
  Place of study: Participants will be recruited from the diabetes clinic, Sohag university hospital.
  Type of the study: Cross-Sectional Comparative study.
  Patients:
  v Study group: participants of the study will meet the following criteria:
  Ø Inclusion criteria:
  ü Age: 30-55 y
  ü Type of diabetes: Type 2
  ü Duration of diabetes: Within 1 Year of diagnosis of Type 2 diabetes mellitus according to World Health Organization 1999 criteria
  ü Gender: Both males & females
  Ø Exclusion criteria:
  Patients who had known conditions that could present with neuropathy such as hereditary sensory neuropathy, vitamin B12 or folate deficiency, paraneoplastic conditions, autoimmune diseases, uremia, hypothyroidism, and ethanol abuse.

SUMMARY:
The study aims to Compare the diagnostic accuracy of the Michigan Neuropathy Screening Instrument (MNSI) (using MNS questionnaire, ,Inspection, vibratory sensation, Ankle reflexes Exam, 10 g monofilament needle examination), routine NCS, and the U/S of the median, posterior tibial, and sural nerves in identifying diabetic peripheral neuropathy in patients recently diagnosed with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* ü Age: 30-55 y

ü Type of diabetes: Type 2

ü Duration of diabetes: Within 1Year of diagnosis of Type 2 diabetes mellitus according to World Health Organization 1999 criteria

Exclusion Criteria:

* Patients who had known conditions that could present with neuropathy such as hereditary sensory neuropathy, vitamin B12 or folate deficiency, paraneoplastic conditions, autoimmune diseases, uremia, hypothyroidism, and ethanol abuse.

Ages: 33 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Place of study: Participants will be recruited from the diabetes clinic, Sohag university hospital.
  * Type of the study: Cross-Sectional Comparative study.
  * Patients:
  v Study group: participants of the study will meet the following criteria:
  Ø Inclusion criteria:
  ü Age: 30-55 y
  ü Type of diabetes: Type 2
  ü Duration of diabetes: Within 1Year of diagnosis of Type 2 diabetes mellitus according to World Health Organization 1999 criteria
  ü Gender: Both males & females
  Ø Exclusion criteria:
  Patients who had known conditions that could present with neuropathy such as hereditary sensory neuropathy, vitamin B12 or folate deficiency, paraneoplastic conditions, autoimmune diseases, uremia, hypothyroidism, and ethanol abuse.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Early detection of Diabetic Neuropathy | Searching in patients diagnosed within 1 year or less
  Utilizing the Michigan Neuropathy Screening Instrument, routine nerve conduction study, and nerve ultrasound for early detection of Diabetic Neuropathy

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medecine Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided